CLINICAL TRIAL: NCT05328687
Title: Examination of Muscle Stiffness, Tenderness and Pressure Pain Thresholds During a Cycle of Botulinum Toxin A Treatment in Chronic Migraine Patients
Acronym: BTACM
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Henrik Schytz, Consultant in Neurology, Danish Headache Center
Other Study IDs: DanishHC180322Botox
Record Dates: First submitted 2022-03-18; First posted 2022-04-14 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Shear wave elastography — or measuring the muscle stiffness, we use a linear 9 MHz ultrasound probe (9L) and the Logic E9 scanner, both from GE Healthcare (Chalfont St Giles, UK). All measurements are performed with the probe parallel to the muscle fibers. We will measure the stiffness of the trapezius muscle in the middle botulinum toxin A injection side (G1) according to the PREEMPT protocol. All data are saved as images by the observer and subsequently analyzed by a blinded observer.

SUMMARY:
Preventive treatment with botulinum toxin A injections is standard care for chronic migraine and follows the PREEMPT protocol. Patients are injected at 31 locations in the frontal, corrugator and procerus muscle, the temporalis muscle, the occipitalis muscle, the cervical paraspinal muscle group and the trapezius muscles (11). The treatment is repeated every 12 weeks, performed by specially trained medical doctors or nurses.

We will measure elastography of the trapezius muscle before and 5-6 weeks after botox injection. In addition measure with QST

DETAILED DESCRIPTION:
Study population

The population considered for inclusion in the study is patients with CM treated with botulinum toxin A injections every third months at DHC. This is an observational study, and inclusion will not affect treatment. Patients will be included consecutively.

Inclusion criteria

Patients being treated (or are starting treatment) with botulinum toxin A injections in the clinical setting at the DHC. Treatment is based on confirmed CM-diagnosis according to the ICHD-III (4), diagnosed by headache specialists at DHC

Aged 18 - 65 years

Able to sign an informed consent

Exclusion criteria

Medication overuse headache

Known cervical disorders, e.g. cervical spine disc prolapses, whiplash or spinal stenosis

Change in other pharmacological preventive medication during the study period. Stable pharmacological preventive medication is allowed.

Treatment with botulinum toxin A injections

Preventive treatment with botulinum toxin A injections is standard care for chronic migraine and follows the PREEMPT protocol. Patients are injected at 31 locations in the frontal, corrugator and procerus muscle, the temporalis muscle, the occipitalis muscle, the cervical paraspinal muscle group and the trapezius muscles (11). The treatment is repeated every 12 weeks, performed by specially trained medical doctors or nurses.

Baseline characteristics

The following information is gathered for research purpose after the patients written consent is obtained.

Information collected from the patient's record or baseline questionnaire at inclusion time

Age, gender, years of migraine and chronic migraine, current use of pharmacological preventive treatment, co-morbidities, number of previous treatments with botulinum toxin A injections, level of physical activity, height (cm) and weight (kg). Any MRI or CT scans of head and neck to verify diagnosis

Information collected from baseline headache and neck pain calendar during 3 months run-in period

Headache days/month, migraine days/month, types of acute medication, days with use of acute medication, days with neck pain and menstrual cycle.

Ultrasound shear-wave elastography

For measuring the muscle stiffness, we use a linear 9 MHz ultrasound probe (9L) and the Logic E9 scanner, both from GE Healthcare (Chalfont St Giles, UK). All measurements are performed with the probe parallel to the muscle fibers. We will measure the stiffness of the trapezius muscle in the middle botulinum toxin A injection side (G1) according to the PREEMPT protocol. All data are saved as images by the observer and subsequently analyzed by a blinded observer.

Total Tenderness Score

Eight paired pericranial muscles and tendons are palpated in a standardized manner with a standardized pressure. small rotating movements are used while palpating. Subjects are asked to rate their tenderness on a 4-point scale (0-3). Scores from each location are added to get a total tenderness score (TTS) ranging from 0 to 48. The eight examined areas are the frontal muscle, temporal muscle, coronoid process, masseter muscle, mastoid process, sternocleidomastoid, trapezius muscle and neck muscle insertions.

Pressure Pain Threshold

Pressure pain threshold will be assessed bilaterally over the temporalis muscle (over injection side G1), the temporalis, and index finger. The pain threshold is defined as the minimal pressure where the sensation of pressure changes to pain. The electronic pressure algometer (Somedic Algometer type 2, Sollentuna, Sweden) will be used. Three PPT measurements are measured over each area with a 30-sec interval between two consecutive measurements at the same area. Pressure will be applied at a rate of 50 kPa /second with a 1 cm2 probe.

ELIGIBILITY:
Inclusion Criteria:

Patients being treated (or are starting treatment) with botulinum toxin A injections in the clinical setting at the DHC. Treatment is based on confirmed CM-diagnosis according to the ICHD-III (4), diagnosed by headache specialists at DHC

Aged 18 - 65 years

Able to sign an informed consent

Exclusion Criteria:

* Medication overuse headache

Known cervical disorders, e.g. cervical spine disc prolapses, whiplash or spinal stenosis

Change in other pharmacological preventive medication during the study period. Stable pharmacological preventive medication is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic migraine referred to the Danish Headache center
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change in muscle stiffness | 6 months
  For measuring the muscle stiffness, we use a linear 9 MHz ultrasound probe (9L) and the Logic E9 scanner, both from GE Healthcare (Chalfont St Giles, UK). All measurements are performed with the probe parallel to the muscle fibers. We will measure the stiffness of the trapezius muscle in the middle botulinum toxin A injection side (G1) according to the PREEMPT protocol. All data are saved as images by the observer and subsequently analyzed by a blinded observer.
Change in total tenderness score | 6 months
  Eight paired pericranial muscles and tendons are palpated in a standardized manner with a standardized pressure. small rotating movements are used while palpating. Subjects are asked to rate their tenderness on a 4-point scale (0-3). Scores from each location are added to get a total tenderness score (TTS) ranging from 0 to 48. The eight examined areas are the frontal muscle, temporal muscle, coronoid process, masseter muscle, mastoid process, sternocleidomastoid, trapezius muscle and neck muscle insertions.
Change in muscle pressure pain threshold | 6 months
  Pressure pain threshold will be assessed bilaterally over the temporalis muscle (over injection side G1), the temporalis, and index finger. The pain threshold is defined as the minimal pressure where the sensation of pressure changes to pain. The electronic pressure algometer (Somedic Algometer type 2, Sollentuna, Sweden) will be used. Three PPT measurements are measured over each area with a 30-sec interval between two consecutive measurements at the same area. Pressure will be applied at a rate of 50 kPa /second with a 1 cm2 probe.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark